CLINICAL TRIAL: NCT02442427
Title: Treatment of Respiratory Syncytial Virus Bronchiolitis in Young Infants With Humanized Monoclonal Antibody: A Randomized Clinical Trial (Palivizumab Study)
Brief Title: "Palivizumab Therapy for RSV-bronchiolitis"
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14302/14
Record Dates: First submitted 2015-05-10; First posted 2015-05-13 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-01

CONDITIONS: Respiratory Syncytial Virus-bronchiolitis
Keywords: Respiratory syncytial virus; Palivizumab; Bronchiolitis; Treatment
MeSH Terms: conditions — Bronchiolitis | interventions — Palivizumab; Antibodies, Monoclonal; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Palivizumab (Active Comparator): A single dose of IV palivizumab
  Interventions: Drug: Palivizumab
- Placebo (Placebo Comparator): An equivalent volume of 0.9% normal saline.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Palivizumab — A single dose of IV palivizumab 15 mg per kilogram body weight (maximum dose =100 mg). The study medication will be given by IV infusion over 30 minutes using a syringe infusion pump.
  Other Names: Monoclonal antibody
  Arms: Palivizumab
Other: Placebo — An equal volume of 0.9% normal saline
  Other Names: 0.9% Normal saline
  Arms: Placebo

SUMMARY:
There is a growing body of literature suggesting that monoclonal antibody could be efficacious in infants with RSV-bronchiolitis, well tolerated with no or clinically insignificant adverse effects.

"The investigators hypothesize that a single dose of iv palivizumab 15 mg/kg in diagnosed infants <3 months old with RSV bronchiolitis will result in fewer infants with readmissions to infirmary/observation or hospital for relapse during 3 weeks of follow-up after discharge".

DETAILED DESCRIPTION:
Setting:

The study will be conducted between September 2014 and April 2018 in the short stay unit of the Pediatric Emergency Center (PEC) of Hamad General Hospital, the only pediatric emergency facility in the State of Qatar. The PEC serves an average of 280 000 patients annually and manages 42 beds in a short stay infirmary unit, to which patients are admitted if they are too ill to be sent home but do not need the intensive care unit. Patients admitted to the unit are assessed at least every 6 hours by a pediatrician to determine readiness for discharge. The length of stay in the unit for bronchiolitis ranges from 6 to 168 hours. In 2012, the investigators saw 8718 infants and young children in 10 666 visits for bronchiolitis. Infants aged ≤3 months presenting to the unit for treatment of viral bronchiolitis will be eligible for the study. Consecutive patients will be recruited except when a study nurse is unavailable or the unit is too busy to recruit.

Procedure:

Patients will be examined on presentation, and those needing additional treatment or observation will be admitted to the short stay infirmary unit. Consecutive patients with bronchiolitis will be assessed for study eligibility within 2 hours. Eligible patients will be enrolled after obtaining written consent. For those who consent, plain chest radiography, and nasopharyngeal swabs will be taken for RSV detection. If the patient has a positive RSV rapid antigen test, patients will be randomized to receive one of the study arms. Bronchiolitis severity score will be measured initially at the start of treatment and then at 12-hour, 24-hour, 36-hour and 48-hour thereafter. The medical team in addition to the parents and patients will be blinded to the medication delivered. Adverse effects in each group will be carefully monitored and documented. Patients will be sent home with salbutamol metered-dose inhalers with an appropriately sized Aerochamber with mask attachment. Daily follow-up by study nurse by telephone is mandatory for 1 week after discharge and then once a week for 2 weeks thereafter. The patient could return to the pediatric emergency center earlier if needed. At all revisits for the same illness, nasopharyngeal swabs will be taken for RSV rapid antigen test and the result recorded.

Study Intervention:

* Active arm: A single dose of IV palivizumab 15 mg per kilogram body weight (maximum dose =100 mg).
* Control arm: Placebo (an equivalent volume of 0.9% normal saline).

ELIGIBILITY:
Inclusion Criteria:

* Infants ≤ 3 months-old, presenting to the main pediatric ER with acute bronchiolitis associated with positive RSV rapid antigen test.

Exclusion Criteria:

* Patients will be excluded from the study if they had 1 or more of the following characteristics:

  * Received monoclonal antibody or IVIG within the last 3 months prior to randomization.
  * Receipt of steroids within 2 days before randomization.
  * Hypersensitivity to monoclonal antibodies or immunoglobulin products.
  * Immunodeficiency.
  * Suspected sepsis.
  * Seizure disorders.
  * Neuromuscular disorders.
  * Congenital heart disease.
  * Major congenital anomalies of respiratory tract.

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 420 (Estimated)
Dates: Start 2014-09; Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Readmission to either infirmary/observation or hospital or PICU during 3 weeks of follow-up after discharge | 3 weeks

SECONDARY OUTCOMES:
Time to medical readiness for discharge | 4 weeks
Revisit to any medical facility for the same illness | 4 weeks
Admission to PICU during initial admission | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Khalid Alansari, Principal Investigator — Hamad Medical Corporation, Doha, Qatar
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alansari K, Toaimah FH, Almatar DH, El Tatawy LA, Davidson BL, Qusad MIM. Monoclonal Antibody Treatment of RSV Bronchiolitis in Young Infants: A Randomized Trial. Pediatrics. 2019 Mar;143(3):e20182308. doi: 10.1542/peds.2018-2308. Epub 2019 Feb 13. PMID 30760509